CLINICAL TRIAL: NCT00345358
Title: Evaluate Immunogenicity, Safety & Reactogenicity of GSK Biologicals' 10-valent Pneumococcal Conjugate Vaccine Given as Catch-up Immunization in Children Older Than 7 mo of Age or as 3-dose Primary Immunization in Children Before 6 mo of Age
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' 10-valent Pneumococcal Conjugate Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 107058
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-07

CONDITIONS: Infections, Streptococcal
Keywords: Booster vaccination; Catch-up vaccination; Pneumococcal vaccine; Immunogenicity; Safety; Pneumococcal disease
MeSH Terms: conditions — Streptococcal Infections; Pneumococcal Infections | interventions — PHiD-CV vaccine; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

ARMS (4):
- Synflorix <6M Group (Active Comparator): This group consisted of subjects up to 6 months of age at first vaccination who received 3 doses of Synflorix™ vaccine co-administered with Infanrix™ IPV/Hib at 3, 4 and 5 months of age and a booster dose of the same vaccines at 12-15 months of age. Vaccines were administrated intramuscularly in the right (Synflorix™) or the left (Infanrix™ IPV/Hib ) thigh or deltoid region (deltoid region only for children >12 months of age if muscle size was adequate).
  Interventions: Biological: Synflorix; Biological: Infanrix IPV/Hib
- Synflorix 7-11M Group (Experimental): This group consisted of subjects 7 to 11 months of age at first vaccination who received 2 doses of Synflorix™, one first dose at enrolment followed by a second dose one month later, and a booster dose at 12-15 months of age. The Synflorix™ vaccine was administrated intramuscularly in the right thigh or deltoid region (deltoid region only for children >12 months of age if muscle size was adequate).
  Interventions: Biological: Synflorix
- Synflorix 12-23M Group (Experimental): This group consisted of subjects 12 to 23 months inclusive at first vaccination who received 2 doses of Synflorix™, one first dose at enrolment followed by a second dose 2 months later. The Synflorix™ vaccine was administrated intramuscularly in the right thigh or deltoid region (deltoid region only for children >12 months of age if muscle size was adequate).
  Interventions: Biological: Synflorix
- Synflorix >=24M Group (Experimental): This group consisted of subjects aged between 24 months (inclusive) to 5 years (inclusive) at vaccination who received one dose of Synflorix™. The Synflorix™ vaccine was administrated intramuscularly in the right thigh or deltoid region (deltoid region only for children >12 months of age if muscle size was adequate).
  Interventions: Biological: Synflorix

INTERVENTIONS:
Biological: Synflorix — 1, 2, 3 or 4 Intramuscular injections, depending on age group
  Other Names: Pneumococcal conjugate vaccine GSK1024850A.
Biological: Infanrix IPV/Hib — 4 intramuscular injections
  Other Names: DTPa-IPV/Hib
  Arms: Synflorix <6M Group

SUMMARY:
The purpose of this phase IIIb study is to determine whether children who have not received a 3-dose primary vaccination with the pneumococcal conjugate vaccine before their 6 months of age, can receive the vaccine as part of a catch-up immunization schedule. The immunogenicity, safety and reactogenicity of GSK Biologicals' pneumococcal conjugate vaccine will be evaluated for four different age groups with different schedules:

< 6 months of age group: 3-dose primary vaccination + a booster dose. 7 to 11 months of age group: 2-dose primary vaccination + a booster dose. 12 to 23 months of age group: 2-dose vaccination; no booster dose. 24 months to 5 years of age group: 1-dose vaccination; no booster dose. Children below 6 months of age will receive concomitantly a DTPa-IPV/Hib vaccine.

DETAILED DESCRIPTION:
The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007

ELIGIBILITY:
Inclusion Criteria:

* Male or female between, and including

  * 9-12 weeks of age at the time of first vaccination for the <6 Mo group.
  * 7-11 months of age at the time of first vaccination for the 7-11 Mo group.
  * 12-23 months of age at the time of first vaccination for the 12-23 Mo group.
  * 24 months to 5 years at the time of first vaccination for the >= 24 Mo group.
* Subjects for whom the investigator believes that their parents/guardians can and will comply with the requirements of the protocol
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Born after a gestation period between 36 and 42 weeks.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the entire study period for each age-group.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting one month before and ending one month after each dose of vaccine(s).
* Previous vaccination against S. pneumoniae.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* History of seizures (this criterion does not apply to subjects who have had a single, uncomplicated febrile convulsion in the past) or neurological disease.
* Acute disease at the time of enrolment.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination
* A family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the entire study period.

Ages: 9 Weeks to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2006-09-18 (Actual); Primary Completion 2007-11-15 (Actual); Study Completion 2007-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Finland (8):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kotka
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Vantaa

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Vesikari T, Karvonen A, Korhonen T, Karppa T, Sadeharju K, Fanic A, Dieussaert I, Schuerman L. Immunogenicity of 10-valent pneumococcal nontypeable Haemophilus Influenzae Protein D Conjugate Vaccine when administered as catch-up vaccination to children 7 months to 5 years of age. Pediatr Infect Dis J. 2011 Aug;30(8):e130-41. doi: 10.1097/INF.0b013e31821d1790. PMID 21540760
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 107058 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107058 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107058 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107058 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107058 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107058 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included a primary (PRI) phase (all groups) and a booster (BST) phase (only 10Pn <6M and Synflorix 7-11M Groups).
Pre-assignment Details: At screening the following was performed: informed consent was obtained from & signed by subjects' parents/guardians, check for inclusion/exclusion criteria and precautions was performed as regards contraindications to vaccination, and medical history of subjects was collected. Subjects' pre-vaccination body temperature was evaluated.
Period: Primary Vaccination Phase
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group | Synflorix 12-23M Group | Synflorix >=24M Group
Started | 150 | 150 | 150 | 150
Completed | 145 | 146 | 142 | 148
Not Completed | 5 | 4 | 8 | 2
Not completed — Other | 0 | 1 | 1 | 0
Not completed — Adverse event, non-fatal | 3 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 4 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2 | 2
Period: Booster Vaccination Phase
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group | Synflorix 12-23M Group | Synflorix >=24M Group
Started | 145 | 145 | 0 | 0
Completed | 141 | 145 | 0 | 0
Not Completed | 4 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group | Synflorix 12-23M Group | Synflorix >=24M Group | Total
Number analyzed (Participants) | 150 | 150 | 150 | 150 | 600
Age, Continuous [Mean (Standard Deviation); unit: Months] | 10.8 (1.09) | 8.3 (1.2) | 17.9 (3.19) | 36.6 (11.87) | 18.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 68 | 76 | 72 | 282
  Male | 84 | 82 | 74 | 78 | 318
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White-Caucasian/European heritage | 149 | 148 | 149 | 149 | 595
  White - Arabic / north African heritage | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or other pacific Islande | 0 | 1 | 0 | 0 | 1
  Other (unspecified) | 0 | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F Antibody Concentrations >= 0.20 Microgram Per Milliliter (µg/mL). (Primary/Full Vaccination)
Description: Anti-pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody concentrations were assessed by 22F-inhibition Enzyme-Linked Immuno-Sorbent Assay (ELISA) method. The >=0.20 microgram per milliliter (microg/mL) cut-off corresponded to the seroprotection cut-off as regards anti-pneumococcal serotypes antibody concentrations. Seropositivity status, defined as anti-pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody concentrations ≥ 0.05 microg/mL.
Time Frame: At one month after primary (Synflorix <6M & Synflorix 7-11M Groups) or after the full (Synflorix 12-23M & Synflorix >=24M Groups) vaccination course with Synflorix™, that is Month (M)3 for Synflorix <6M & 12-23M groups, M2 for Synflorix 7-11M Group, & M1
Population: The analysis was performed on the Primary According-To-Protocol cohort for immunogenicity,which included all evaluable subjects with immunogenicity data available.This included subjects with assay results available for antibodies against at least one study vaccine antigen component and at least one bloodsampling time point after primary vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group | Synflorix 12-23M Group | Synflorix >=24M Group
Number analyzed (Participants) | 131 | 135 | 133 | 140
Participants
  Anti-1 | 128 | 135 | 132 | 135
  Anti-4 | 128 | 135 | 133 | 140
  Anti-5: number analyzed (Participants) | 131 | 135 | 133 | 138
  Anti-5 | 130 | 134 | 131 | 135
  Anti-6B | 95 | 69 | 108 | 96
  Anti-7F | 130 | 135 | 133 | 140
  Anti-9V | 128 | 129 | 130 | 132
  Anti-14: number analyzed (Participants) | 131 | 135 | 133 | 139
  Anti-14 | 130 | 132 | 132 | 127
  Anti-18C | 127 | 135 | 133 | 140
  Anti-19F | 122 | 129 | 131 | 140
  Anti-23F: number analyzed (Participants) | 131 | 135 | 133 | 139
  Anti-23F | 114 | 95 | 122 | 93

2. Secondary Outcome: Antibody Concentrations Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. (Primary/Full Vaccination)
Description: Antibodies assessed for this outcome measure were those against the vaccine pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (ANTI-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F). Antibody concentrations were measured by 22F enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). Seropositivity = Anti-pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody concentrations ≥0.05 µg/mL.
Time Frame: At 1 month after the administration of the primary (< 6 months and 7-11 months groups) or the full (12-23 months and >= 24 months groups) vaccination course, with Synflorix™ vaccine.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group | Synflorix 12-23M Group | Synflorix >=24M Group
Number analyzed (Participants) | 131 | 135 | 133 | 140
μg/mL
  Anti-1 | 1.2 [1.02 to 1.42] | 1.19 [1.05 to 1.35] | 1.22 [1.06 to 1.4] | 0.77 [0.66 to 0.89]
  Anti-4 | 1.84 [1.57 to 2.15] | 3.47 [3.03 to 3.97] | 4.21 [3.77 to 4.69] | 5.72 [5 to 6.54]
  Anti-5: number analyzed (Participants) | 131 | 135 | 133 | 138
  Anti-5 | 2.04 [1.75 to 2.37] | 1.72 [1.51 to 1.96] | 1.8 [1.57 to 2.06] | 1.16 [0.99 to 1.36]
  Anti-6B | 0.37 [0.29 to 0.48] | 0.21 [0.16 to 0.26] | 0.53 [0.43 to 0.65] | 0.38 [0.3 to 0.47]
  Anti-7F | 2.03 [1.76 to 2.33] | 2.1 [1.83 to 2.41] | 3.62 [3.22 to 4.06] | 2.6 [2.25 to 3.01]
  Anti-9V | 1.33 [1.14 to 1.55] | 0.91 [0.78 to 1.07] | 1.5 [1.3 to 1.73] | 1.01 [0.84 to 1.22]
  Anti-14: number analyzed (Participants) | 131 | 135 | 133 | 139
  Anti-14 | 3 [2.61 to 3.46] | 2.3 [1.95 to 2.72] | 4.24 [3.64 to 4.95] | 1.36 [1.06 to 1.74]
  Anti-18C | 1.84 [1.5 to 2.26] | 4.82 [4.14 to 5.61] | 9.2 [8.22 to 10.29] | 4.65 [4.06 to 5.31]
  Anti-19F | 1.61 [1.28 to 2.02] | 3.36 [2.68 to 4.2] | 5.45 [4.63 to 6.41] | 5.26 [4.34 to 6.39]
  Anti-23F: number analyzed (Participants) | 131 | 135 | 133 | 139
  Anti-23F | 0.62 [0.5 to 0.76] | 0.4 [0.32 to 0.5] | 0.88 [0.73 to 1.05] | 0.37 [0.3 to 0.47]

3. Secondary Outcome: Antibody Concentrations Against Pneumococcal Cross-reactive Serotypes 6A and 19A. (Primary/Full Vaccination)
Description: Antibodies assessed for this outcome measure were those against the vaccine pneumococcal serotypes 6A, 19A (ANTI-6A, -19A). Antibody concentrations were measured by 22F enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). Seropositivity = Anti-pneumococcal cross-reactive serotypes 6A and 19A antibody concentrations ≥ 0.05 µg/mL.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group | Synflorix 12-23M Group | Synflorix >=24M Group
Number analyzed (Participants) | 132 | 135 | 133 | 138
μg/mL
  Anti-6A | 0.1 [0.08 to 0.12] | 0.06 [0.05 to 0.08] | 0.23 [0.18 to 0.29] | 0.24 [0.19 to 0.31]
  Anti-19A: number analyzed (Participants) | 131 | 135 | 133 | 138
  Anti-19A | 0.09 [0.07 to 0.11] | 0.12 [0.1 to 0.15] | 0.86 [0.71 to 1.05] | 0.65 [0.53 to 082]

4. Secondary Outcome: Opsonophagocytic Activity Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. (Primary/Full Vaccination)
Description: OPA titers against pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Opsono-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F) were calculated, expressed as geometric mean titers (GMTs) and tabulated. Seropositivity = Opsonophagocytic activity against pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F >= 8. Antibody titers < 8 were given an arbitrary value of half the cut-off for the purpose of GMT calculation.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group | Synflorix 12-23M Group | Synflorix >=24M Group
Number analyzed (Participants) | 44 | 48 | 51 | 41
Titers
  Opsono-1 | 17.3 [10.9 to 27.5] | 14.8 [9.3 to 23.6] | 14.2 [9 to 22.4] | 17.5 [9.4 to 32.3]
  Opsono-4: number analyzed (Participants) | 41 | 46 | 50 | 36
  Opsono-4 | 675.6 [475.4 to 960] | 524 [361.8 to 758.9] | 912.1 [617.8 to 1346.8] | 2227.6 [1694 to 2929.3]
  Opsono-5: number analyzed (Participants) | 42 | 46 | 50 | 39
  Opsono-5 | 52.6 [33.7 to 82.2] | 33.7 [21.4 to 53.3] | 47.5 [30.2 to 74.8] | 14.1 [9.1 to 22]
  Opsono-6B: number analyzed (Participants) | 38 | 45 | 49 | 34
  Opsono-6B | 296 [130.3 to 672.2] | 25.4 [11.1 to 58.4] | 304.3 [143.8 to 644.2] | 331.7 [99.1 to 1109.8]
  Opsono-7F: number analyzed (Participants) | 43 | 46 | 48 | 38
  Opsono-7F | 1775.1 [1057.8 to 2978.8] | 2342.5 [1555.2 to 3528.2] | 4164.2 [2840.4 to 6105] | 3282.2 [2105.1 to 5117.6]
  Opsono-9V: number analyzed (Participants) | 41 | 44 | 50 | 37
  Opsono-9V | 1281.1 [895 to 1833.7] | 2209.6 [1628.6 to 2997.8] | 3525.8 [2675.4 to 4646.4] | 4526 [3581.7 to 5719.3]
  Opsono-14: number analyzed (Participants) | 42 | 48 | 51 | 40
  Opsono-14 | 1523.3 [1028.7 to 2255.6] | 1818.9 [1356.4 to 2439.2] | 2277.2 [1804.9 to 2873] | 1957.4 [1516.6 to 2526.3]
  Opsono-18C: number analyzed (Participants) | 41 | 46 | 51 | 38
  Opsono-18C | 181.8 [120.8 to 273.5] | 971.7 [723.2 to 1305.5] | 1765.3 [1330.5 to 2342.2] | 2051.4 [1558.3 to 2700.5]
  Opsono-19F: number analyzed (Participants) | 42 | 43 | 50 | 41
  Opsono-19F | 194.7 [101.7 to 372.7] | 225.6 [128.6 to 395.7] | 592.7 [367.3 to 956.4] | 634.3 [400.2 to 1005.4]
  Opsono-23F: number analyzed (Participants) | 41 | 45 | 49 | 41
  Opsono-23F | 925.8 [422.6 to 2028.3] | 561.1 [273.7 to 1150.4] | 1656.4 [1063.6 to 2579.6] | 1575.2 [802.6 to 3091.7]

5. Secondary Outcome: Opsonophagocytic Activity Against Pneumococcal Cross-reactive Serotypes 6A and 19A. (Primary/Full Vaccination)
Description: OPA titers against pneumococcal serotypes 6A, 19A (Opsono-6A, 19A) were calculated, expressed as geometric mean titers (GMTs) and tabulated. Opsonophagocytic activity against cross-reactive pneumococcal serotypes 6A and 19A >= 8. Antibody titers < 8 were given an arbitrary value of half the cut-off for the purpose of GMT calculation.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group | Synflorix 12-23M Group | Synflorix >=24M Group
Number analyzed (Participants) | 43 | 45 | 50 | 38
Titers
  Opsono-6A: number analyzed (Participants) | 41 | 44 | 50 | 35
  Opsono-6A | 14.4 [7.5 to 27.6] | 39.1 [19 to 80.6] | 150.7 [80.7 to 281.3] | 324.6 [142.6 to 738.6]
  Opsono-19: number analyzed (Participants) | 43 | 45 | 49 | 38
  Opsono-19 | 5.1 [3.9 to 6.6] | 6.1 [4.2 to 8.8] | 39.5 [19 to 81.9] | 31.8 [14.3 to 70.7]

6. Secondary Outcome: Antibody Concentrations Against Protein D (Anti-PD). (Primary/Full Vaccination)
Description: Anti-protein D (Anti-PD) antibody concentrations by Enzyme-Linked Immunosorbent Assay (ELISA) were calculated, expressed as geometric mean concentrations (GMCs) in ELISA unit per milli-liter (EL.U/mL) and tabulated. Seropositivity = Anti-PD antibody concentrations >= 100 EL.U/mL. Antibody concentrations < 100 EL.U/mL were given an arbitrary value of half the cut-off for the purpose of GMC calculation.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group | Synflorix 12-23M Group | Synflorix >=24M Group
Number analyzed (Participants) | 131 | 135 | 133 | 139
EL.U/mL | 1637.7 [1430.9 to 1874.3] | 654.2 [577.7 to 741] | 660 [554.9 to 785.1] | 224.8 [185.2 to 272.7]

7. Secondary Outcome: Anti-pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F Antibody Concentrations >= 0.20 µg/mL. (Booster Vaccination)
Description: Anti-pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody concentrations were assessed by 22F-inhibition Enzyme-Linked Immuno-Sorbent Assay (ELISA) method. The >=0.20 microgram per millilitre (microg/mL) cut-off corresponded to the seroprotection cut-off as regards anti-pneumococcal serotypes antibody concentrations. Seropositivity = Anti-pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody concentrations ≥0.05 µg/mL.
Time Frame: Before and one month after the booster dose with Synflorix™ for the < 6 months and 7-11 months groups
Population: The analysis was performed on the Booster According-To-Protocol(ATP) cohort for immunogenicity,which included all evaluable subjects with immunogenicity data available(subjects from the Synflorix <6M & 7-11M groups for whom assay results were available for antibodies against at least one study vaccine antigen component after the booster vaccination
Measure: Number; unit: Subjects
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group
Number analyzed (Participants) | 140 | 114
Subjects
  Anti-1, PRE | 101 | 102
  Anti-1, POST: number analyzed (Participants) | 137 | 114
  Anti-1, POST | 137 | 114
  Anti-4, PRE | 119 | 112
  Anti-4, POST: number analyzed (Participants) | 137 | 114
  Anti-4, POST | 137 | 114
  Anti-5, PRE | 123 | 110
  Anti-5, POST: number analyzed (Participants) | 137 | 114
  Anti-5, POST | 136 | 114
  Anti-6B, PRE | 108 | 97
  Anti-6B, POST: number analyzed (Participants) | 137 | 114
  Anti-6B, POST | 132 | 110
  Anti-7F, PRE | 132 | 114
  Anti-7F, POST: number analyzed (Participants) | 137 | 114
  Anti-7F, POST | 137 | 114
  Anti-9V, PRE | 131 | 108
  Anti-9V, POST: number analyzed (Participants) | 137 | 114
  Anti-9V, POST | 137 | 114
  Anti-14, PRE | 131 | 113
  Anti-14, POST: number analyzed (Participants) | 137 | 114
  Anti-14, POST | 137 | 114
  Anti-18C, PRE | 127 | 114
  Anti-18C, POST: number analyzed (Participants) | 137 | 114
  Anti-18C, POST | 137 | 114
  Anti-19F, PRE | 114 | 112
  Anti-19F, POST: number analyzed (Participants) | 137 | 114
  Anti-19F, POST | 134 | 112
  Anti-23F, PRE | 116 | 98
  Anti-23F, POST: number analyzed (Participants) | 137 | 114
  Anti-23F, POST | 136 | 110

8. Secondary Outcome: Anti-pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F Antibody Concentrations. (Booster Vaccination)
Description: Anti-pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody concentrations were assessed by 22F-inhibition Enzyme-Linked Immuno-Sorbent Assay (ELISA) method. The >=0.20 microgram per millilitre (microg/mL) cut-off corresponded to the seroprotection cut-off as regards anti-pneumococcal serotypes antibody concentrations. Seropositivity status, defined as Anti-pneumococcal serotypes antibody concentrations >=0.05 µg/mL.
Time Frame: Before and one month after the booster dose with Synflorix™ for the < 6 months and 7-11 months groups
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group
Number analyzed (Participants) | 140 | 141
μg/mL
  Anti-1, PRE | 0.29 [0.25 to 0.34] | 0.49 [0.43 to 0.57]
  Anti-1, POST: number analyzed (Participants) | 137 | 141
  Anti-1, POST | 1.84 [1.59 to 2.12] | 1.77 [1.55 to 2.02]
  Anti-4, PRE | 0.56 [0.48 to 0.66] | 1.35 [1.17 to 1.57]
  Anti-4, POST: number analyzed (Participants) | 137 | 141
  Anti-4, POST | 2.98 [2.6 to 3.42] | 3.79 [3.27 to 4.4]
  Anti-5, PRE | 0.51 [0.44 to 0.59] | 0.8 [0.7 to 0.93]
  Anti-5, POST: number analyzed (Participants) | 137 | 141
  Anti-5, POST | 2.21 [1.94 to 2.53] | 2.88 [2.48 to 3.34]
  Anti-6B, PRE | 0.41 [0.34 to 0.5] | 0.48 [0.4 to 0.58]
  Anti-6B, POST: number analyzed (Participants) | 137 | 141
  Anti-6B, POST | 1.62 [1.35 to 1.94] | 1.39 [1.14 to 1.69]
  Anti-7F, PRE | 0.82 [0.72 to 0.94] | 1.58 [1.39 to 1.8]
  Anti-7F, POST: number analyzed (Participants) | 137 | 141
  Anti-7F, POST | 3.31 [2.92 to 3.74] | 3.73 [3.24 to 4.28]
  Anti-9V, PRE | 0.85 [0.73 to 0.98] | 0.79 [0.67 to 0.93]
  Anti-9V, POST: number analyzed (Participants) | 137 | 141
  Anti-9V, POST | 3.41 [2.96 to 3.92] | 2.13 [1.82 to 2.5]
  Anti-14, PRE | 1.03 [0.85 to 1.25] | 2.3 [1.97 to 2.68]
  Anti-14, POST: number analyzed (Participants) | 137 | 141
  Anti-14, POST | 3.96 [3.39 to 4.62] | 5.41 [4.71 to 6.22]
  Anti-18C, PRE | 0.62 [0.53 to 0.74] | 2.58 [2.2 to 3.04]
  Anti-18C, POST: number analyzed (Participants) | 137 | 141
  Anti-18C, POST | 5.28 [4.55 to 6.12] | 9.4 [8.04 to 10.98]
  Anti-19F, PRE | 0.55 [0.44 to 0.7] | 1.99 [1.65 to 2.4]
  Anti-19F, POST: number analyzed (Participants) | 137 | 141
  Anti-19F, POST | 3.38 [2.81 to 4.06] | 5.71 [4.68 to 6.97]
  Anti-23F, PRE | 0.48 [0.39 to 0.58] | 0.57 [0.46 to 0.7]
  Anti-23F, POST: number analyzed (Participants) | 137 | 141
  Anti-23F, POST | 2.76 [2.37 to 3.21] | 1.65 [1.33 to 2.03]

9. Secondary Outcome: Antibody Concentrations Against Pneumococcal Cross-reactive Serotypes 6A and 19A.(Booster Vaccination)
Description: Antibodies assessed for this outcome measure were those against the vaccine pneumococcal serotypes 6A, 19A (ANTI-6A, -19A). Antibody concentrations were measured by 22F enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL).Seropositivity = Anti-pneumococcal cross-reactive serotypes 6A and 19A antibody concentrations ≥ 0.05 μg/mL.
Time Frame: Before and one month after the booster dose with Synflorix™ for the < 6 months and 7-11 months groups
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group
Number analyzed (Participants) | 140 | 114
μg/mL
  Anti-6A, PRE | 0.15 [0.12 to 0.19] | 0.18 [0.14 to 0.23]
  Anti-6A, POST: number analyzed (Participants) | 137 | 114
  Anti-6A, POST | 0.52 [0.4 to 0.68] | 0.55 [0.42 to 0.73]
  Anti-19A, PRE | 0.1 [0.09 to 0.13] | 0.26 [0.21 to 0.32]
  Anti-19A, POST: number analyzed (Participants) | 137 | 114
  Anti-19A, POST | 0.49 [0.39 to 0.61] | 0.99 [0.78 to 1.25]

10. Secondary Outcome: Opsonophagocytic Activity Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. (Booster Vaccination)
Description: OPA titers against pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Opsono-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F) were calculated, expressed as geometric mean titers (GMTs) and tabulated. Seropositivity status, defined as Opsonophagocytic activity against pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F >= 8. Antibody titers < 8 were given an arbitrary value of half the cut-off for the purpose of GMT calculation.
Time Frame: Before and one month after the booster dose with Synflorix™ for the < 6 months and 7-11 months groups
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group
Number analyzed (Participants) | 51 | 40
Titers
  Opsono-1, PRE: number analyzed (Participants) | 51 | 38
  Opsono-1, PRE | 6 [4.5 to 8.1] | 9.9 [5.8 to 16.9]
  Opsono-1, POST: number analyzed (Participants) | 48 | 40
  Opsono-1, POST | 188 [103.6 to 342.5] | 234.1 [127.4 to 430.2]
  Opsono-4, PRE: number analyzed (Participants) | 45 | 37
  Opsono-4, PRE | 22.2 [12.4 to 39.9] | 94 [47.7 to 185.2]
  Opsono-4, POST: number analyzed (Participants) | 48 | 38
  Opsono-4, POST | 1486.3 [1138 to 1941] | 978.3 [720.6 to 1328.1]
  Opsono-5, PRE: number analyzed (Participants) | 48 | 37
  Opsono-5, PRE | 16 [11.1 to 23.1] | 25.8 [16.3 to 41]
  Opsono-5, POST: number analyzed (Participants) | 47 | 39
  Opsono-5, POST | 143.8 [93.6 to 221] | 243 [151.6 to 389.7]
  Opsono-6B, PRE: number analyzed (Participants) | 45 | 31
  Opsono-6B, PRE | 59.3 [29.3 to 120.1] | 122.7 [50.3 to 299.5]
  Opsono-6B, POST: number analyzed (Participants) | 45 | 40
  Opsono-6B, POST | 262 [130.3 to 526.5] | 620.3 [356.5 to 1079.4]
  Opsono-7F, PRE: number analyzed (Participants) | 49 | 33
  Opsono-7F, PRE | 819.6 [451.8 to 1423.8] | 1380.6 [730.3 to 2609.9]
  Opsono-7F, POST: number analyzed (Participants) | 48 | 40
  Opsono-7F, POST | 4199.1 [3364.6 to 5240.6] | 3726.8 [2759.4 to 5033.3]
  Opsono-9V, PRE: number analyzed (Participants) | 50 | 37
  Opsono-9V, PRE | 328.2 [245.4 to 438.8] | 1427 [972.7 to 2093.4]
  Opsono-9V, POST: number analyzed (Participants) | 48 | 38
  Opsono-9V, POST | 2198 [1718.6 to 2811.1] | 2241.2 [1758.7 to 2856]
  Opsono-14, PRE: number analyzed (Participants) | 46 | 37
  Opsono-14, PRE | 158.6 [82.6 to 304.6] | 883.8 [597.9 to 1306.2]
  Opsono-14, POST: number analyzed (Participants) | 48 | 40
  Opsono-14, POST | 2224.7 [1674.1 to 2956.5] | 1859.4 [1452.1 to 2380.9]
  Opsono-18C, PRE: number analyzed (Participants) | 42 | 33
  Opsono-18C, PRE | 6.5 [4.2 to 10] | 395.9 [219.9 to 712.8]
  Opsono-18C, POST: number analyzed (Participants) | 48 | 38
  Opsono-18C, POST | 650.3 [437.4 to 966.8] | 1332.9 [926.3 to 1918]
  Opsono-19F, PRE: number analyzed (Participants) | 49 | 38
  Opsono-19F, PRE | 18.7 [12 to 29.3] | 43.3 [23.3 to 80.4]
  Opsono-19F, POST: number analyzed (Participants) | 47 | 38
  Opsono-19F, POST | 418.4 [237.8 to 736.4] | 513.1 [265.8 to 990.2]
  Opsono-23F, PRE: number analyzed (Participants) | 49 | 34
  Opsono-23F, PRE | 700.6 [376.5 to 1303.9] | 675.8 [293.2 to 1557.4]
  Opsono-23F, POST: number analyzed (Participants) | 48 | 40
  Opsono-23F, POST | 3594.5 [2676.8 to 4826.8] | 1770 [1148.4 to 2728]

11. Secondary Outcome: Opsonophagocytic Activity Against Pneumococcal Cross-reactive Serotypes 6A and 19A. (Booster Vaccination)
Description: as for outcome 5
Time Frame: Before and one month after the booster dose with Synflorix™ for the < 6 months and 7-11 months groups
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group
Number analyzed (Participants) | 47 | 37
Titers
  Opsono-6A, PRE: number analyzed (Participants) | 41 | 33
  Opsono-6A, PRE | 31.9 [15.9 to 63.9] | 140.1 [69.2 to 283.3]
  Opsono-6A, POST: number analyzed (Participants) | 43 | 36
  Opsono-6A, POST | 188.6 [96.9 to 367] | 302.2 [168.7 to 541.5]
  Opsono-19A, PRE: number analyzed (Participants) | 47 | 35
  Opsono-19A, PRE | 5.7 [4.2 to 7.7] | 7 [3.9 to 12.6]
  Opsono-19A, POST: number analyzed (Participants) | 44 | 37
  Opsono-19A, POST | 16.1 [8.6 to 30.1] | 36.8 [16.2 to 83.8]

12. Secondary Outcome: Antibody Concentrations Against Protein D. (Booster Vaccination)
Description: as for outcome 6
Time Frame: Before and one month after the booster dose with Synflorix™ for the < 6 months and 7-11 months groups
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group
Number analyzed (Participants) | 140 | 114
EL.U/mL
  Anti-PD, PRE | 750.4 [631.2 to 892] | 563.2 [475.5 to 666.9]
  Anti-PD, POST: number analyzed (Participants) | 135 | 114
  Anti-PD, POST | 2900.7 [2481.5 to 3390.8] | 1942 [1614.5 to 2335.9]

13. Secondary Outcome: Anti-diphtheria (Anti-D) and Anti-tetanus Toxoids (Anti-T) Antibody Concentrations. (Primary Vaccination)
Description: Concentrations of antibodies are presented as geometric mean concentrations expressed as International units per milliliter (IU/mL). Seroprotection status, defined as: Anti-D & anti-T antibody concentrations >=0.1 IU/mL. Since only "Synflorix <6M Group" had received DTPa-IPV/Hib, therefore only that group was assessed for this Outcome.
Time Frame: At 1 month after the administration of the primary vaccination course (Month [M]3 = POST-PRY) with Infanrix™ IPV/Hib vaccine when co-administered with Synflorix™, for the < 6 months Group.
Population: The analysis was performed on the Primary ATP cohort for immunogenicity, which included all evaluable subjects with immunogenicity data available for at least one study vaccine antigen component and at least one time point after primary vaccination. Only Synflorix <6M Group received DTPa-IPV/Hib, thus only that group was assessed for this Outcome.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Synflorix <6M Group
Number analyzed (Participants) | 132
IU/mL
  Anti-D, POST-PRY: number analyzed (Participants) | 131
  Anti-D, POST-PRY | 0.961 [0.813 to 1.137]
  Anti-T, POST-PRY | 2.38 [2.131 to 2.659]

14. Secondary Outcome: Anti-polyribosyl Ribitol Phosphate (PRP) Antibody Concentrations. (Primary Vaccination)
Description: Concentrations of antibodies are presented as geometric mean concentrations expressed as micrograms per milliliter (µg/mL). Seroprotection status, defined as: anti-PRP antibody concentrations >=0.15 µg/mL and >= 1.0 µg/mL. Since only "Synflorix <6M Group" had received DTPa-IPV/Hib, therefore only that group was assessed for this Outcome.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix <6M Group
Number analyzed (Participants) | 132
μg/mL | 2.886 [2.305 to 3.615]

15. Secondary Outcome: Anti-pertussis Toxoid (PT), Anti-filamentous Haemagglutinin (FHA) and Anti-pertactin (PRN) Antibody Concentrations. (Primary Vaccination)
Description: Concentrations of antibodies are presented as geometric mean concentrations expressed as enzyme-linked immunosorbent assay (ELISA) unit per milliliter (EL.U/mL). Seropositivity status, defined as: Anti-PT, anti-FHA & anti-PRN antibody concentrations >= 5 EL.U/mL. Since only "Synflorix <6M Group" had received DTPa-IPV/Hib, therefore only that group was assessed for this Outcome.
Time Frame: At 1 month after the administration of the primary vaccination course(Month [M]3 = POST-PRY) with Infanrix™ IPV/Hib vaccine when co-administered with Synflorix™, for the < 6 months Group
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix <6M Group
Number analyzed (Participants) | 130
EL.U/mL
  Anti-PT, POST-PRY: number analyzed (Participants) | 129
  Anti-PT, POST-PRY | 51.5 [46.5 to 57]
  Anti-FHA, POST-PRY: number analyzed (Participants) | 127
  Anti-FHA, POST-PRY | 211.4 [192.7 to 231.8]
  Anti-PRN, POST-PRY | 103.2 [90.7 to 117.4]

16. Secondary Outcome: Anti-polio Type 1, 2 and 3 Titers. (Primary Vaccination)
Description: Titers of antibodies are presented as geometric mean titers. Seroprotection status, defined as: Anti-polio type 1/2/3 titers >= 8.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix <6M Group
Number analyzed (Participants) | 17
Titers
  Anti-Polio 1, POST-PRY | 55.5 [30 to 102.6]
  Anti-Polio 2, POST-PRY: number analyzed (Participants) | 16
  Anti-Polio 2, POST-PRY | 20.2 [9.7 to 41.9]
  Anti-Polio 3, POST-PRY: number analyzed (Participants) | 16
  Anti-Polio 3, POST-PRY | 162.3 [73.5 to 358.5]

17. Secondary Outcome: Booster Vaccine Response to PT, FHA and PRN
Description: Booster vaccine response to PT, FHA and PRN, defined as appearance of antibodies in subjects who were seronegative (S-) prior to the booster dose (i.e., with concentrations < 5 EL.U/mL), and at least two-fold increase of pre-booster vaccination antibody concentrations in those who were seropositive (S+) prior to the booster dose (i.e., with concentrations >= 5 EL.U/ mL). Since only "Synflorix <6M Group" had received DTPa-IPV/Hib, therefore only that group was assessed for this Outcome.
Time Frame: Before and one month after the booster dose with Synflorix™
Population: The analysis was performed on the Booster ATP cohort for immunogenicity, which included all evaluable subjects (from Synflorix <6M & 7-11M groups) for whom assay results were available for at least one study vaccine antigen after the booster vaccination. Only Synflorix <6M Group received DTPa-IPV/Hib, only that group was assessed for this Outcome.
Measure: Number; unit: Subjects
Arm/Group | Synflorix <6M Group
Number analyzed (Participants) | 136
Subjects
  Anti-PT-Pre-booster status S-: number analyzed (Participants) | 14
  Anti-PT-Pre-booster status S- | 14
  Anti-PT-Pre-booster status S+: number analyzed (Participants) | 121
  Anti-PT-Pre-booster status S+ | 117
  Anti-FHA-Pre-booster status S-: number analyzed (Participants) | 0
  Anti-FHA-Pre-booster status S+ | 131
  Anti-PRN-Pre-booster status S-: number analyzed (Participants) | 12
  Anti-PRN-Pre-booster status S- | 12
  Anti-PRN-Pre-booster status S+: number analyzed (Participants) | 124
  Anti-PRN-Pre-booster status S+ | 123

18. Secondary Outcome: Number of Subjects Solicited Local Symptoms (Any and Grade 3). (Primary Vaccination)
Description: Assessed local symptoms were pain, redness and swelling. Any = Occurrence of the specified solicited local symptom, regardless of intensity. Grade 3 Pain = Crying when limb was moved/spontaneously painful. Grade 3 Redness/Swelling = Redness/swelling at injection site larger than (>) 30 millimeters (mm). Across doses= across the 3 doses (D1, D2 and D3) of the Synflorix™ vaccine co-administered with Infranrix™ in the <6 months priming group; across the 2 doses of the Synflorix™ vaccine in the 7-11 months priming group; across the 2 doses of the Synflorix™ vaccine in the 12-23 months priming group and in the 1 dose of Synflorix™ vaccine in the ≥24 months priming group.
Time Frame: Within 4-day (Days 0-3) following the primary vaccination
Population: The analysis was performed on the Primary Total Vaccinated cohort, which included all vaccinated subjects (e.g. all subjects who received at least one primary dose).
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group | Synflorix 12-23M Group | Synflorix >=24M Group
Number analyzed (Participants) | 149 | 148 | 149 | 148
Participants
  Any Pain, D1 | 63 | 52 | 93 | 102
  Grade 3 Pain, D1 | 10 | 5 | 21 | 24
  Any Redness, D1 | 60 | 83 | 57 | 65
  Grade 3 Redness, D1 | 3 | 9 | 3 | 9
  Any Swelling, D1 | 37 | 48 | 39 | 32
  Grade 3 Swelling, D1 | 5 | 10 | 6 | 7
  Any Pain, D2: number analyzed (Participants) | 146 | 147 | 143 | 0
  Any Pain, D2 | 51 | 41 | 84 | 0
  Grade 3 Pain, D2: number analyzed (Participants) | 146 | 147 | 143 | 0
  Grade 3 Pain, D2 | 0 | 0 | 12 | 0
  Any Redness, D2: number analyzed (Participants) | 146 | 147 | 143 | 0
  Any Redness, D2 | 66 | 70 | 52 | 0
  Grade 3 Redness, D2: number analyzed (Participants) | 146 | 147 | 143 | 0
  Grade 3 Redness, D2 | 0 | 4 | 2 | 0
  Any Swelling, D2: number analyzed (Participants) | 146 | 147 | 143 | 0
  Any Swelling, D2 | 38 | 39 | 38 | 0
  Grade 3 Swelling, D2: number analyzed (Participants) | 146 | 147 | 143 | 0
  Grade 3 Swelling, D2 | 2 | 6 | 7 | 0
  Any Pain, D3: number analyzed (Participants) | 145 | 0 | 0 | 0
  Any Pain, D3 | 40 | 0 | 0 | 0
  Grade 3 Pain, D3: number analyzed (Participants) | 145 | 0 | 0 | 0
  Grade 3 Pain, D3 | 3 | 0 | 0 | 0
  Any Redness, D3: number analyzed (Participants) | 145 | 0 | 0 | 0
  Any Redness, D3 | 58 | 0 | 0 | 0
  Grade 3 Redness, D3: number analyzed (Participants) | 145 | 148 | 149 | 148
  Grade 3 Redness, D3 | 1 | 0 | 0 | 0
  Any Swelling, D3: number analyzed (Participants) | 145 | 0 | 0 | 0
  Any Swelling, D3 | 33 | 0 | 0 | 0
  Grade 3 Swelling, D3: number analyzed (Participants) | 145 | 0 | 0 | 0
  Grade 3 Swelling, D3 | 2 | 0 | 0 | 0
  Any Pain, Across | 89 | 63 | 113 | 102
  Grade 3 Pain, Across | 13 | 5 | 29 | 24
  Any Redness, Across | 90 | 95 | 79 | 65
  Grade 3 Redness, Across | 4 | 12 | 4 | 9
  Any Swelling, Across | 68 | 66 | 59 | 32
  Grade 3 Swelling, Across | 9 | 14 | 12 | 7

19. Secondary Outcome: Number of Subjects With Solicited Local Symptoms (Any and Grade 3). (Booster Vaccination)
Description: Assessed local symptoms were pain, redness and swelling. Any = Occurrence of the specified solicited local symptom, regardless of intensity. Grade 3 Pain = Crying when limb was moved/spontaneously painful. Grade 3 Redness/Swelling = Redness/swelling at injection site larger than (>) 30 millimeters (mm).
Time Frame: Within 4-day (Days 0-3) following the booster vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group
Number analyzed (Participants) | 144 | 145
Participants
  Any Pain | 91 | 64
  Grade 3 Pain | 11 | 3
  Any Redness | 80 | 73
  Grade 3 Redness | 11 | 5
  Any Swelling | 55 | 45
  Grade 3 Swelling | 10 | 7

20. Secondary Outcome: Number of Subjects With Solicited General Symptoms (Any and Grade 3). (Booster Vaccination)
Description: Assessed solicited general symptoms were Drowsiness, Irritability, Loss of appetite (Loss Appet.) and Fever (rectal temperature higher than [≥] 38.0 degrees Celsius [°C]),. Any = Occurrence of the specified solicited general symptom, regardless of intensity or relationship to vaccination. Grade 3 Drowsiness = Drowsiness that prevented normal activity. Grade 3 Irr./Fuss. = Crying that could not be comforted/prevented normal activity. Grade 3 Loss of appetite = Subject did not eat at all. Grade 3 Fever = Rectal temperature higher than (>) 40.0°C.
Time Frame: Within 4 day (Days 0-3) following the booster vacination
Population: The analysis was performed on the Booster Total Vaccinated, which cohort included all subjects from the Synflorix <6M & Synflorix 7-11M groups months groups, who received the booster dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group
Number analyzed (Participants) | 144 | 145
Participants
  Any Drowsiness | 73 | 57
  Grade 3 Drowsiness | 3 | 3
  Any Fever (Rectally) | 63 | 33
  Grade 3 Fever (Rectally) | 1 | 0
  Any Irritability | 109 | 71
  Grade 3 Irritability | 5 | 3
  Any Loss of Appet. | 57 | 35
  Grade 3 Loss of Appet. | 1 | 3

21. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs). (Primary Vaccination)
Description: An unsolicited AE was defined as any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For the marketed products administered in the study, this also included failure to produce expected benefits (i.e. lack of efficacy), abuse or misuse of the product. Any = Occurrence of an unsolicited AE, regardless of intensity or relationship to vaccination.
Time Frame: Within 31-day (Days 0-30) post primary vaccination
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group | Synflorix 12-23M Group | Synflorix >=24M Group
Number analyzed (Participants) | 150 | 150 | 150 | 150
Participants | 100 | 116 | 101 | 54

22. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs). (Booster Vaccination)
Description: as for outcome 21
Time Frame: Within 31 day (Days 0-30) following the booster vaccination
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group
Number analyzed (Participants) | 145 | 145
Participants | 90 | 63

23. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) (Primary Vaccination)
Description: A SAE was defined as any medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity in a subject. AE(s) considered as SAE(s) also included invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that did not result in hospitalisation, as per the medical or scientific judgement of the physician. Any = Occurrence of a SAE, regardless of relationship to vaccination.
Time Frame: During the Primary vaccination course up until start of Booster vaccination course
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group | Synflorix 12-23M Group | Synflorix >=24M Group
Number analyzed (Participants) | 150 | 150 | 150 | 150
Participants | 17 | 5 | 2 | 0

24. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs). (Booster Vaccination)
Description: as for outcome 23
Time Frame: During the booster vaccination course
Population: The analysis was performed on the Booster Total Vaccinated, which cohort included all subjects from the Synflorix <6M & Synflorix 7-11M groups, who received the booster dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group
Number analyzed (Participants) | 145 | 145
Participants | 1 | 1

25. Secondary Outcome: Number of Subjects With Solicited General Symptoms (Primary Vaccination)
Description: Assessed solicited general symptoms were Drowsiness, Irritability, Loss of appetite (Loss Appet.) and Fever (rectal temperature higher than [≥] 38.0 degrees Celsius [°C]),. Any = Occurrence of the specified solicited general symptom, regardless of intensity or relationship to vaccination. Grade 3 Drowsiness = Drowsiness that prevented normal activity. Grade 3 Irr./Fuss. = Crying that could not be comforted/prevented normal activity. Grade 3 Loss of appetite = Subject did not eat at all. Grade 3 Fever = Rectal temperature higher than (>) 40.0°C. Across doses= across the 3 doses (D1, D2 and D3) of the Synflorix™ vaccine co-administered with Infranrix™ in the <6 months priming group; across the 2 doses of the Synflorix™ vaccine in the 7-11 months priming group; across the 2 doses of the Synflorix™ vaccine in the 12-23 months priming group and in the 1 dose of Synflorix™ vaccine in the ≥24 months priming group.
Time Frame: Within 4-day (Days 0-3) following the primary vaccination
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group | Synflorix 12-23M Group | Synflorix >=24M Group
Number analyzed (Participants) | 149 | 148 | 149 | 148
Participants
  Drowsiness, Dose 1 | 101 | 70 | 63 | 55
  Grade 3 Drowsiness, Dose 1 | 2 | 1 | 1 | 1
  Any Fever (Rectally), Dose 1 | 54 | 34 | 30 | 10
  Grade 3 Fever (Rectally), Dose 1 | 0 | 0 | 0 | 0
  Any Irritability, Dose 1 | 122 | 90 | 90 | 62
  Grade 3 Irritability, Dose 1 | 12 | 5 | 4 | 2
  Any Loss of Appet, Dose 1 | 45 | 42 | 46 | 41
  Grade 3 Loss of Appet., Dose 1 | 0 | 0 | 3 | 0
  Any Drowsiness, Dose 2: number analyzed (Participants) | 146 | 147 | 143 | 0
  Any Drowsiness, Dose 2 | 64 | 51 | 48 | 0
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 146 | 147 | 143 | 0
  Grade 3 Drowsiness, Dose 2 | 0 | 0 | 2 | 0
  Any Fever (Rectally), Dose 2: number analyzed (Participants) | 146 | 147 | 143 | 0
  Any Fever (Rectally), Dose 2 | 60 | 34 | 24 | 0
  Grade 3 Fever (Rectally), Dose 2: number analyzed (Participants) | 146 | 147 | 143 | 0
  Grade 3 Fever (Rectally), Dose 2 | 0 | 0 | 0 | 0
  Any Irritability, Dose 2: number analyzed (Participants) | 146 | 147 | 143 | 0
  Any Irritability, Dose 2 | 103 | 78 | 62 | 0
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 146 | 147 | 143 | 0
  Grade 3 Irritability, Dose 2 | 2 | 0 | 3 | 0
  Any Loss of Appet., Dose 2: number analyzed (Participants) | 146 | 147 | 143 | 0
  Any Loss of Appet., Dose 2 | 31 | 35 | 31 | 0
  Grade 3 Loss of Appet., Dose 2: number analyzed (Participants) | 146 | 147 | 143 | 0
  Grade 3 Loss of Appet., Dose 2 | 0 | 0 | 1 | 0
  Any Drowsiness, Dose 3: number analyzed (Participants) | 145 | 0 | 0 | 0
  Any Drowsiness, Dose 3 | 53 | 0 | 0 | 0
  Grade 3 Drowsiness, Dose 3: number analyzed (Participants) | 145 | 0 | 0 | 0
  Grade 3 Drowsiness, Dose 3 | 0 | 0 | 0 | 0
  Any Fever (Rectally), Dose 3: number analyzed (Participants) | 145 | 0 | 0 | 0
  Any Fever (Rectally), Dose 3 | 40 | 0 | 0 | 0
  Grade 3 Fever (Rectally), Dose 3: number analyzed (Participants) | 145 | 0 | 0 | 0
  Grade 3 Fever (Rectally), Dose 3 | 0 | 0 | 0 | 0
  Any Irritability, Dose 3: number analyzed (Participants) | 145 | 0 | 0 | 0
  Any Irritability, Dose 3 | 83 | 0 | 0 | 0
  Grade 3 Irritability, Dose 3: number analyzed (Participants) | 145 | 0 | 0 | 0
  Grade 3 Irritability, Dose 3 | 3 | 0 | 0 | 0
  Any Loss of Appet., Dose 3: number analyzed (Participants) | 145 | 0 | 0 | 0
  Any Loss of Appet., Dose 3 | 22 | 0 | 0 | 0
  Grade 3 Loss of Appet., Dose 3: number analyzed (Participants) | 145 | 0 | 0 | 0
  Grade 3 Loss of Appet., Dose 3 | 0 | 0 | 0 | 0
  Any Drowsiness, Across | 122 | 92 | 90 | 55
  Grade 3 Drowsiness, Across | 2 | 1 | 3 | 1
  Any Fever (Rectally), Across | 95 | 55 | 47 | 10
  Grade 3 Fever (Rectally),Across | 0 | 0 | 0 | 0
  Any Irritability, Across | 143 | 112 | 107 | 62
  Grade 3 Irritability, Across | 70 | 62 | 62 | 41
  Grade 3 Loss of Appet., Across | 0 | 0 | 4 | 0

26. Secondary Outcome: Anti-diphtheria (Anti-D) and Anti-tetanus Toxoids (Anti-T) Antibody Concentrations.(Booster Vaccination)
Description: Concentrations of antibodies are presented as geometric mean concentrations expressed as International units per milliliter (IU/mL). Seroprotection status, defined as: Anti-D & anti-T antibody concentrations >= 0.1 IU/mL.. Since only "Synflorix <6M Group" had received DTPa-IPV/Hib, therefore only that group was assessed for this Outcome.
Time Frame: Before (M9 = PRE-BST) and one month after the booster dose (M10 = POST-BST) with Infanrix™ IPV/Hib vaccine when co-administered with Synflorix™, for the < 6 months Group.
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Synflorix <6M Group
Number analyzed (Participants) | 140
IU/mL
  Anti-D, PRE-BST | 0.218 [0.185 to 0.258]
  Anti-D, POST-BST: number analyzed (Participants) | 137
  Anti-D, POST-BST | 4.093 [3.578 to 4.683]
  Anti-T, PRE-BST | 0.708 [0.616 to 0.813]
  Anti-T, POST-BST: number analyzed (Participants) | 137
  Anti-T, POST-BST | 10.245 [9.302 to 11.283]

27. Secondary Outcome: Anti-polyribosyl Ribitol Phosphate (PRP) Antibody Concentrations. (Booster Vaccination)
Description: Concentrations of antibodies are presented as geometric mean concentrations expressed as micrograms per milliliter (µg/mL). Seroprotection status, defined as: anti-PRP antibody concentrations >= 0.15 µg/mL and >= 1.0 µg/mL. Since only "Synflorix <6M Group" had received DTPa-IPV/Hib, therefore only that group was assessed for this Outcome.
Time Frame: as for outcome 26
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix <6M Group
Number analyzed (Participants) | 140
μg/mL
  Anti-PRP, PRE-BST | 0.458 [0.366 to 0.573]
  Anti-PRP, POST-BST: number analyzed (Participants) | 136
  Anti-PRP, POST-BST | 21.244 [16.778 to 26.9]

28. Secondary Outcome: Anti-pertussis Toxoid (PT), Anti-filamentous Haemagglutinin (FHA) and Anti-pertactin (PRN) Antibody Concentrations. (Booster Vaccination)
Description: Concentrations of antibodies are presented as geometric mean concentrations expressed as enzyme-linked immunosorbent assay (ELISA) unit per milliliter (EL.U/mL). Seropositivity status, defined as: Anti-PT, anti-FHA & anti-PRN antibody concentrations >=5 EL.U/mL. Since only "Synflorix <6M Group" had received DTPa-IPV/Hib, therefore only that group was assessed for this Outcome.
Time Frame: as for outcome 26
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix <6M Group
Number analyzed (Participants) | 140
EL.U/mL
  Anti-PT, PRE-BST | 11.2 [9.8 to 12.7]
  Anti-PT, POST-BST: number analyzed (Participants) | 136
  Anti-PT, POST-BST | 88.6 [79.5 to 98.7]
  Anti-FHA, PRE-BST | 49.2 [43.3 to 55.9]
  Anti-FHA, POST-BST: number analyzed (Participants) | 137
  Anti-FHA, POST-BST | 407.1 [368.5 to 449.8]
  Anti-PRN, PRE-BST | 17.2 [14.7 to 20.1]
  Anti-PRN, POST-BST: number analyzed (Participants) | 137
  Anti-PRN, POST-BST | 276.6 [240.9 to 317.6]

29. Secondary Outcome: Titers of Antibodies Against Polio Type 1, 2 and 3 (Anti-polio 1, 2 and 3). (Booster Vaccination)
Description: Titers of antibodies are presented as geometric mean titers. Seroprotection status, defined as: Anti-polio type 1/2/3 titers >= 8. Since only "Synflorix <6M Group" had received DTPa-IPV/Hib, therefore only that group was assessed for this Outcome.
Time Frame: as for outcome 26
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix <6M Group
Number analyzed (Participants) | 140
Titers
  Anti-Polio 1, PRE--BST: number analyzed (Participants) | 16
  Anti-Polio 1, PRE--BST | 19.1 [10.4 to 34.9]
  Anti-Polio 1, POST-BST: number analyzed (Participants) | 13
  Anti-Polio 1, POST-BST | 617 [302.3 to 1259.2]
  Anti-Polio 2, PRE-BST: number analyzed (Participants) | 18
  Anti-Polio 2, PRE-BST | 14 [7.6 to 25.7]
  Anti-Polio 2, POST-BST: number analyzed (Participants) | 13
  Anti-Polio 2, POST-BST | 498.5 [198.1 to 1254.3]
  Anti-Polio 3, PRE-BST: number analyzed (Participants) | 18
  Anti-Polio 3, PRE-BST | 20.1 [10.6 to 38.2]
  Anti-Polio 3, POST-BST: number analyzed (Participants) | 13
  Anti-Polio 3, POST-BST | 1234.1 [688.3 to 2212.4]

ADVERSE EVENTS:
Time Frame: Solicited & Unsolicited AEs: During the 4 & 31 days post PRI/BST vaccination; SAEs: during PRI and BST Phases.
Description: Note that: 1) For Synflorix™ <6M Group & Synflorix 7-11M Group SAEs were reported during both PRI and BST Phases 2) The BST Phase safety follow-up is not applicable for the Synflorix™ 12-23M Group & Synflorix >=24M Group, as no booster doses were administered.
Arm/Group | Synflorix <6M Group | Synflorix 7-11M Group | Synflorix 12-23M Group | Synflorix >=24M Group
Serious Adverse Events (participants affected / at risk) | 18/150 | 6/150 | 2/150 | 0/150
Other Adverse Events (participants affected / at risk) | 149/150 | 145/150 | 144/150 | 135/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Synflorix <6M Group (N=150) | Synflorix 7-11M Group (N=150) | Synflorix 12-23M Group (N=150) | Synflorix >=24M Group (N=150)
Bronchitis chronic - PRI (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Psychomotor retardation - PRI (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper - PRI (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia - PRI (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Pyelonephritis acute - PRI (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis - PRI (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis rotavirus - PRI (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Otitis media - PRI (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Exanthema subitum - PRI (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza - PRI (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis - PRI (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection - PRI (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection - BST (Infections and infestations) | 1/145 (1) | 0/145 (0) | 0/0 (0) | 0/0 (0)
Gastroenteritis - BST (Infections and infestations) | 0/145 (0) | 1/145 (1) | 0/0 (0) | 0/0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Synflorix <6M Group (N=150) | Synflorix 7-11M Group (N=150) | Synflorix 12-23M Group (N=150) | Synflorix >=24M Group (N=150)
Conjunctivitis (Eye disorders) | 7 (7) | 13 (13) | 4 (4) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 20 (22) | 20 (24) | 5 (6)
Decreased appetite (Metabolism and nutrition disorders) | 94 (155) | 74 (112) | 62 (77) | 41 (42)
Diarrhoea (Gastrointestinal disorders) | 11 (12) | 16 (21) | 14 (15) | 5 (5)
Ear infection (Infections and infestations) | 0 (0) | 15 (18) | 3 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 109 (266) | 109 (232) | 79 (112) | 65 (66)
Injection site haematoma (General disorders) | 9 (9) | 5 (5) | 0 (0) | 2 (2)
Injection site induration (General disorders) | 16 (22) | 12 (14) | 12 (15) | 1 (1)
Irritability (Psychiatric disorders) | 145 (426) | 124 (241) | 107 (152) | 63 (64)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 11 (14) | 0 (0)
Otitis media (Infections and infestations) | 19 (20) | 28 (34) | 20 (23) | 10 (11)
Pain (General disorders) | 114 (245) | 90 (157) | 113 (177) | 102 (103)
Pyrexia (General disorders) | 120 (238) | 87 (138) | 60 (74) | 19 (19)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) | 5 (5) | 4 (4) | 1 (1)
Rhinitis (Infections and infestations) | 37 (52) | 33 (47) | 18 (22) | 4 (4)
Somnolence (Nervous system disorders) | 130 (291) | 103 (178) | 90 (111) | 56 (57)
Swelling (General disorders) | 88 (163) | 77 (132) | 59 (77) | 32 (32)
Teething (Gastrointestinal disorders) | 14 (17) | 22 (28) | 4 (5) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 60 (80) | 43 (59) | 21 (24) | 7 (8)
Vomiting (Gastrointestinal disorders) | 8 (8) | 9 (9) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.